CLINICAL TRIAL: NCT05946720
Title: Aggression From the Perspective of Patients and Nurses: An Integrated Study on the Evaluation of Aggression in Psychiatric Clinics
Brief Title: Aggression From the Perspective of Patients and Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, SEDA TEK SEVİNDİK, Ph.D, RN, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 117
Record Dates: First submitted 2023-06-23; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Aggression
Keywords: aggression; aggression in psychiatry clinics; perception of aggression; risk level of violence
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Intervention Model Description: pre- post test, training and control group, randomise controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taining group (Experimental): Nurses in the training group were given training on aggression and the use of BVC.
  Interventions: Other: Training including aggression and the use of BVC.
- Control group (No Intervention): Nurses in the control group were not trained, till the study ends.

INTERVENTIONS:
Other: Training including aggression and the use of BVC. — After obtaining verbal consent from the nurses who met the inclusion criteria of the study before the pre-test was applied to the nurses, the nurses who volunteered to participate in the study were randomized within their own clinic using the simple randomization method. For this, after the data collection form was distributed before the pre-test, the nurses were asked to write the letter that came to them on the data collection form and not forget it. In order for nurses to be included in the training or comparison group, the letter A, written on the closed papers in the box prepared for simple randomization, represents the Education group, and the letter B represents the comparison group.
  Arms: Taining group

SUMMARY:
The research, was planned in a randomized controlled design, aiming to evaluate the effect of the training given to nurses working in psychiatric clinics on the use of aggression and BVC (Broset Violence Checklist) on the nurses' perceptions of aggression and the compliance of the use of BVC, which they evaluated for the patients watched in the videos, with the BVC determined by expert opinion.

The study was conducted in Adana Doctor Ekrem Tok Mental Health and Diseases Hospital between July 2021 and April 2022. A total of 97 nurses working in psychiatric clinics, 47 in the training group and 50 in the comparison group, participated in the study. A pre-test was administered to the nurses and nurses in the training group were randomized and given training including aggression and BVC use. After the training, a post-test was administered to all nurses.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* To have been working in the hospital where the research was conducted for at least 1 year,
* To have no vision, hearing and speech problems.

Exclusion Criteria:

* To want to withdraw from the research at any stage of the research,
* Not completing or not being able to complete the research for any reason,
* To work in the filiation team during the research process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Perception of Aggression Scale | Procedure (one week before the training)
  The scale has a 5-point Likert-type rating system ranging from strongly disagree (1) to strongly agree (5) and consists of 29 items. The items have two subscales: functional (functional - acceptable / healthy response) and dysfunctional (dysfunctional - unacceptable / undesirable aggression). For each subscale, the average of the relevant item scores will be calculated.
Broset Violence Checklist | Procedure (one week before the training and one day after the training)
  A score of "1" is given in the presence of each item of the BVC, and "0" in the absence of it. In the next evaluations of the patient, if there is an increase in the relevant item compared to the previous one, the behavior score is scored as "1", the habitual or same level behavior is considered absent and scored as "0". If there is no more in the case of a patient with a flood than before, the relevant item score should be "0". If an increase in the level of exuberance is observed, it should be scored as "1". After the six items are scored in this way, the evaluation is made over the total score. A total score of "0" indicates that the patient has a low severity risk level. "1- 2 points" indicates moderate risk of violence and necessitates measures to prevent violence. "3-6 points" refers to a high risk of violence.
Perception of Aggression Scale | Procedure (one day after the training)
  The scale has a 5-point Likert-type rating system ranging from strongly disagree (1) to strongly agree (5) and consists of 29 items. The items have two subscales: functional (functional - acceptable / healthy response) and dysfunctional (dysfunctional - unacceptable / undesirable aggression). For each subscale, the average of the relevant item scores will be calculated.
Broset Violence Checklist | Procedure (one day after the training)
  A score of "1" is given in the presence of each item of the BVC, and "0" in the absence of it. In the next evaluations of the patient, if there is an increase in the relevant item compared to the previous one, the behavior score is scored as "1", the habitual or same level behavior is considered absent and scored as "0". If there is no more in the case of a patient with a flood than before, the relevant item score should be "0". If an increase in the level of exuberance is observed, it should be scored as "1". After the six items are scored in this way, the evaluation is made over the total score. A total score of "0" indicates that the patient has a low severity risk level. "1- 2 points" indicates moderate risk of violence and necessitates measures to prevent violence. "3-6 points" refers to a high risk of violence.

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova Üniversitesi, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No